CLINICAL TRIAL: NCT01610999
Title: Pilot Study of Lymphoid Tumor Microenvironmental Dysruption Prior to Autologous Stem Cell Transplantation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unavailability of study article
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Plerixafor
Record Dates: First submitted 2012-03-16; First posted 2012-06-04 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Chronic Lymphocytic Leukemia; Lymphoma; Multiple Myeloma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma; Multiple Myeloma | interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): 0.24 mg/kg plerixafor on day 1
  Interventions: Drug: Plerixafor
- Cohort B (Experimental): 0.24 mg/kg plerixafor daily on days 1 & 2
  Interventions: Drug: Plerixafor
- Cohort C (No Intervention): Six "control" subjects will have research bloods drawn but receive no plerixafor.

INTERVENTIONS:
Drug: Plerixafor — Plerixafor will be dosed according to actual body weight. Each dose will be capped at 24 mg (single vial). Plerixafor will be administered subcutaneously according to the assigned cohort starting two hours before the scheduled start of high dose chemotherapy.
  Other Names: Mozobil
  Arms: Cohort A; Cohort B

SUMMARY:
In order to keep our immune systems healthy over our lifetime, certain cells in the bone marrow and lymph nodes called stromal cells nurture the immune cells and protect them from damage. Stromal cells and blood cells communicate using a protein called SDF1a. The investigators think that cancer cells including lymphoma and multiple myeloma can trick the stromal cells into helping them avoid damage from chemotherapy by using SDF1a.

Plerixafor is a drug developed to block the effects of SDF1a and has been approved by the Federal Drug Administration (FDA) for use in humans to help release blood stem cells from the bone marrow for use in transplantation. The use of plerixafor to interrupt communication between stromal cells and cancer has not been approved by the FDA and is experimental.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Subjects must have documented, relapsed/refractory or high-risk primary lymphoid malignancy
* Subjects must have evidence of residual disease prior to transplant, but need not have measurable or strictly evaluable disease
* Subjects must be eligible candidates for high dose chemotherapy with either BEAM or single-agent melphalan preparative regimens and autologous stem cell transplantation at Tufts Medical Center (See Appendix B for anticipated transplant schedules)
* Subjects must be able to provide informed consent to the research procedure

Exclusion Criteria:

* Uncontrolled infection
* Active heart disease as evidenced by myocardial infarction within 6 months, uncontrolled arrhythmia, or angina.
* Creatinine clearance estimated < 50 ml/min.
* HIV infection or evidence of active chronic hepatitis
* Unable or unwilling to comply with required study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The rate of grade 2 or greater adverse events related to study participation will be compared to historical controls matched for diagnosis and chemotherapy regimen. | 2 hours before high dose chemotherapy
  Confirm the safety of the addition of plerixafor as a single dose or as a two-day dose commencing 2 hours before the high dose chemotherapy regimen prior to autologous stem cell transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas K Klein, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No